CLINICAL TRIAL: NCT04406077
Title: The Use of Ligasure (r) for Cutting and Coagulations of Tissues in Hydrocelectomy Surgery
Brief Title: The Use of Ligasure (r) for Hydrocelectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0117-17-HYMC
Record Dates: First submitted 2020-05-06; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Hydrocele
MeSH Terms: conditions — Testicular Hydrocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients suffering from hydrocele, underwent treatment using Ligasure device.
  Interventions: Device: Ligasure

INTERVENTIONS:
Device: Ligasure — Using ligasure to treat hydrocele

SUMMARY:
Hydrocele is a condition of fluid retention around the testes, which causes swallowing, pain, with interfering with the normal testes function. however, during activity, this can interfere with everyday activity (running, sexual intercourse). The treatment for hydrocele I surgical. The study aim to test the safety and efficacy of the Ligasure (r) device for cutting and coagulating tissues during hydrocelectomy.

DETAILED DESCRIPTION:
Hydrocele is a condition of fluid retention around the testes, which causes swallowing, pain, with interfering with the normal testes function. however, during activity, this can interfere with everyday activity (running, sexual intercourse). The treatment for hydrocele I surgical. The study aim to test the safety and efficacy of the Ligasure (r) device for cutting and coagulating tissues during hydrocelectomy. during the study, males, 18 - 81 who suffer from hydrocele underwent hydrocelectomy using Ligasure (20 cm) without using sutures.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 81 males
* Diagnosed with unilateral hydrocele

Exclusion Criteria:

* Bilateral hydrocele
* infected hydrocele
* hydrocele secondary to tumor

Ages: 18 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
resolution of hydrocele | Three weeks after the surgery
  The patients will undergo full urological physical exam to screen for signs of hydrocele. The testes size and manual palpation will be included in the assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No